CLINICAL TRIAL: NCT01112332
Title: : Use of an Innovative Weight-bearing Measuring Device to Determine Normative Percentage Body-Weight/Weight-Bearing Values and Weight-bearing Gait Characteristics in Different Physiologic Conditions
Brief Title: Weight-bearing Measuring Device to Determine Normative Percentage Body-Weight/Weight-Bearing Values and Weight-bearing Gait Characteristics
Acronym: SSW001
Status: Available | Type: Expanded Access
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 042-2010
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Percentage Body-Weight; Weight-Bearing Values; Weight-bearing Gait Characteristics

INTERVENTIONS:
Device: SmartStep insole — Smart StepTM is an innovative biofeedback and monitoring system designed to help clinicians effectively guide patients with compromised lower limb function due to orthopedic or neurological trauma towards optimal gait performance. It records and analyzes key gait parameters and provides instantaneous and accurate audio and visual feedback.

SUMMARY:
The objective of this clinical trial is to determine normative Percentage Body-Weight/Weight-Bearing Values and Weight-bearing Gait Characteristics in different physiologic conditions

1. Values in increasing speeds from walking to running.
2. Changing resistance and incline on an elliptical trainer
3. Ground jogging.
4. Stair climbing.
5. Treadmill running.
6. Walking.

DETAILED DESCRIPTION:
Background information Orthopedic surgeons and rehabilitation physicians frequently request limited weight-bearing for prolonged periods following certain bony or soft tissue pathologies as well as certain lower - limb surgical procedures. Walking, stair climbing, jogging, elliptical training and running on treadmill are a common activity that the injured athlete will seek to return to as soon as possible following injury or surgery. In order for the physician to be able to advise regarding weight-bearing, the Percentage Body-Weight/Weight-Bearing (PBW/WB) values in increasing walking, jogging speeds, elliptical training must be known. These parameters as well as the gait distribution changes have eluded the rehabilitation community, mainly due to the technical inability to measure these paradigms.

Accurate percentage body weight/weight-bearing (PBW/WB) value analysis in walking has up been investigated in laboratory settings, using balance plate systems and force plate platforms. The aim of this study is to evaluate normal gait characteristics and PBW/WB values using a relatively new hand-held, portable, weight-bearing measuring device (Smartstep™).

During their regular training the participants will use the flexible, light weight, force-sensing insole for few minutes to receive the parameters

1. subjects. In order to accurately control the speed changes, the test measurements will be conducted on a treadmill (Technogym™ "run excite 700"). The tested speeds will be 4,6,8,10,12,14,16,18 and 20 km/hr consecutively. Each subject will run for a 15 second time period for each speed.
2. 25 subjects. The test measurements will be conducted on an Elliptical trainer (Precor USA 576i EFX). The protocol includes 3 tests. In the first test, resistance and incline will be paired together in increasing order at the set device levels of 1, 5, 10, 15, and 20. In the second test, the resistance will be held constant at level 1, while the incline will be increased from levels 1 to 20 in increments of five. In the third test, the incline will remain constant at level 1, while the resistance will be increased from levels 1 to 20 in increments of five. Each subject will be tested over a 20 second time period for each of the changed resistances and inclines. The subjects will be instructed to keep a steady pace within the range of steps/min = 70-95.
3. 40 subjects. The test subjects will be instructed to jog at their normal speed on a solid ground surface over a distance of 16 meters.
4. 40 subjects. The test measurements will be conducted on a flight of 10 stairs, each 17cm high. The subjects will be instructed to ascend and descend the stairs at their normal pace.
5. 40 subjects. The tested speed will be held at 8.5 km/hr on a treadmill (Technogym™ "run excite 700"). Each subject will run for a 15 second time period.
6. 40 subjects. The test subjects will be instructed to walk at their normal speed on a solid ground surface over a distance of 16 meters.

The results will be analyzed and a table of normal values will be established including average PBW/WB values for the entire, hind and fore-foot as well as gait distribution changes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients more than 18 years old, that usually training in Lerner Central Sport, Hebrew University - Jerusalem
* Pain free in their hip, knee and ankle/foot joints for at least a 3 month period prior to testing
* Patients who are willing to participate in the trial, to come to all scheduled visits and to sign the informed consent forms.

Exclusion Criteria:

* Patients receiving other methods of treatment to this area,
* Patients with concomitant other injury of the hip, knee, ankle or foot.
* Previous surgery in the hip, knee, ankle/foot less than 2 years previously.
* Non cooperative patient with the basic rehab program.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2010-03

CONTACTS AND LOCATIONS:
Overall Officials: Ezequiel Palmanovich, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Jerusalem Sports Medicine Institute, Lerner Sports Center, Hebrew University of Jerusalem, Jerusalem, Israel